CLINICAL TRIAL: NCT00924209
Title: Phase II Study of Neoadjuvant Gemcitabine, Cisplatin and Bevacizumab in Stage IIIA (N2), Non-Squamous Cell Non-Small Cell Lung Cancer
Brief Title: A Phase II Study of Neo-Adjuvant Gemcitabine, Cisplatin and Bevacizumab in Stage IIIA (N2) Non-Squamous Cell Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Caryn Steakley, R.N., Deputy Clinical Director, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090107; 09-C-0107; NCT00874081 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: NSCLC; Stage IIIA (N2)
Keywords: Neoadjuvant; Stage IIIA (N2); Cisplatin; Gemcitabine; Bevacizumab; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Bevacizumab; Surgical Procedures, Operative; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stage IIIA lung cancer patients (Experimental): Non-squamous cell non small cell lung cancer treated with 1250 mg/m^2 gemcitabine dose for two doses on day 1 and day 8 every 21 days,80 mg/m^2 cisplatin day 1 every 21 days for 3 cycles, 7.5 mg/kg bevacizumab on day 1 every 21 days for first 2 cycles only, and 100 mg/m^2 intravenous, and 100 mg/m^2 etoposide intravenous per day for consecutive 3 days on days 1 to 3 every 3 weeks for 4 cycles.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Bevacizumab; Procedure: Surgery; Drug: Etoposide

INTERVENTIONS:
Drug: Gemcitabine — 1250 mg/m^2 dose for two doses on days 1 and 8
  Other Names: Gemzar
Drug: Cisplatin — 80 mg/m^2 on day 1
  Other Names: Cisplatinum
Drug: Bevacizumab — 7.5 mg/m^2 on day 1 every 21 days for first two cycles only
  Other Names: Avastin
Procedure: Surgery — thoracotomy with lobectomy/pneumonectomy and mediastinal lymph node dissection 4-6 weeks post completion of last cycle of cisplatin
Drug: Etoposide — 100 mg/m^2 intravenous per day for consecutive 3 days on days 1 to 3 every 3 weeks for 4 cycles.
  Other Names: Vepesid

SUMMARY:
Background:

* Surgical resection is the treatment of choice for patients with lung cancer, and cure after resection generally depends on whether lymph nodes are involved. A patient with Stage IIIA (N2) lung cancer has cancer in the lymph nodes involving the center of the chest (mediastinum).
* Studies have shown that surgery alone as a treatment for Stage IIIA (N2) lung cancer is not as effective as chemotherapy followed by surgery.
* Giving chemotherapy upfront may prevent the spread of Stage IIIA (N2) lung cancer tumors, and may shrink the tumors to allow adequate surgery to be performed. It is also thought that chemotherapy is usually better tolerated before major surgery than after, so higher doses can be given.

Objectives:

* To determine the effectiveness of the combination of three anti-cancer drugs (gemcitabine, cisplatin, and bevacizumab) given before surgery.
* To find out what effects this drug combination may have on the patient and the cancer.
* To determine if the combination of all three drugs given prior to surgery is more effective and as safe, safer, or less safe than other drug combinations given before surgery.

Eligibility:

* Patients with Stage IIIA (N2) lung cancer who have not had chemotherapy, radiation, or surgery to treat the cancer.

Design:

* Evaluations before the treatment period to determine eligibility:
* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Tests to evaluate heart and lung function, such as an echocardiogram.
* Blood and urine tests.
* Disease evaluation with computed tomography (CT), chest X-ray, positron emission tomography (PET) scans, and bronchoscopy/mediastinoscopy (examinations of the inside of the chest and lungs).
* Treatment with intravenous gemcitabine, cisplatin, and bevacizumab for three 21-day cycles.
* Cycles 1 and 2 - Gemcitabine on day 1 and day 8, cisplatin on day 1, bevacizumab on day 1.
* Cycle 3 - Gemcitabine on day 1 and day 8, cisplatin on day 1 (no bevacizumab).
* Physical examinations and tests will be conducted throughout each cycle.
* Surgery will take place 4 to 6 weeks after the last cycle if heart and lung functions are satisfactory and if the cancer remains stable.
* Chemotherapy (four 21-day cycles of cisplatin and etoposide treatments), further evaluations and examinations, and followup studies will take place 4 to 8 weeks after the surgery.

DETAILED DESCRIPTION:
Background:

* Stage IIIA-N2 is considered one of the most therapeutically challenging and controversial subsets of lung cancer. This heterogenous group of patients have tumors which range from minimal N2 (found incidentally during or after surgery) to multi-station bulky N2 disease. The extent of mediastinal involvement has an inverse correlation with survival.
* The 5-year survival ranges from 5-8% in patients with bulky N2 disease, to nearly 35% in patients with single station, microscopic N2 involvement.
* Neo-adjuvant chemotherapy and chemo-radiotherapy have been shown to be superior to surgery alone.
* Platinum-based induction chemotherapy in early and locally advanced non small cell lung cancer (NSCLC) results in a radiological down-staging in at least 50% of patients, and a pathological complete response rate of approximately 5%.
* Concurrent chemo-radiotherapy as an induction regimen increases the radiological and pathological down-staging rate, but at the cost of increasing the morbidity and mortality of a surgical intervention.
* Expectations have now turned towards a possible incremental effect of adding a targeted biological agent to a standard induction treatment.

Primary Objectives:

* To determine the safety of neo-adjuvant Gemcitabine/Cisplatin and Bevacizumab in stage IIIA-N2 non small cell lung cancer (NSCLC)
* To determine the pathological complete response rate
* To determine the resectability rate
* To determine the extent of surgery

Eligibility:

* Histologically confirmed stage IIIA-N2 NSCLC (non-squamous)
* No previous chemotherapy, radiotherapy, surgery or biological therapy for lung cancer
* Adequate organ and bone marrow function

Design:

* Multi-center, international (United States Of America (USA)/Croatia), open labeled phase II trial
* Following a Simon two-stage optimal design

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically documented non squamous cell non-small cell lung cancer and confirmed by the pathological laboratories at participating centers.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than 20 mm with conventional techniques or as greater than 10 mm with spiral computed tomography (CT) scan.
* Stage IIIA (N2) disease. All patients will require a baseline mediastinoscopy to ensure histological proof of N2 disease.
* No prior treatment for lung cancer including chemotherapy, radiotherapy, surgery or biological therapy.
* Age greater than or equal to 18 years (males or non-pregnant females).
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky greater than 60 percent).
* Adequate pulmonary and cardiovascular function to tolerate planned surgical resection:

  * Pulmonary Function criteria:

    * Partial pressure of oxygen (paO2) greater than 65 mmHg, partial pressure of carbon dioxide (paCO2) less than 45 mmHg on room air arterial blood gas (ABG).
    * Anticipated post-op forced expiratory volume 1 (FEV1) greater than or equal to 40 percent predicted.
    * Anticipated post-op carbon monoxide diffusing capacity (DLCO) greater than or equal to 40 percent predicted.
    * If anticipated post-op FEV1 or DLCO less than percent predicted, must have volume of oxygen (VO2) greater than 15ml/kg on oxygen consumption study.
  * Cardiac criteria:

    * Left ventricular ejection fraction (LVEF) greater than 40 percent.
    * No pulmonary hypertension or right ventricular (RV) dysfunction.
    * No unstable angina.
* Serum Creatinine less than or equal to 1.5mg/dl
* Hemoglobin (baseline) greater than or equal to 10.0g/dl
* Absolute neutrophil count greater than or equal to 1,500/m^3 and platelets greater than or equal to 100,000/m^3.
* aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times the upper limit of normal (ULN), total bilirubin less than or equal to 1.5 times the ULN (In patients with evidence of Gilberts disease, elevated bilirubin should not be related to tumor or other liver diseases and should be less than or equal 2 times the upper limit of normal).
* The ability to understand and the willingness to sign a written informed consent document and the ability to comply with the requirements of the protocol.
* Women of childbearing potential must have a negative pregnancy test and both men and women must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

EXCLUSION CRITERIA:

* Squamous cell cancer or mixed tumors with small cell elements.
* Tumor of any histology in close proximity to a major vessel or cavitation. (Any tumor abutting an interlobar, main pulmonary artery, vena cava or major vein will be excluded).
* History of hemoptysis (bright red blood of one-half teaspoon or more [greater than or equal to 2.5 mL] unrelated to any diagnostic procedure. (Patients who have a history of hemoptysis that occurred greater than 3 months prior to study entry and that is assessed not to be related to tumor may be eligible).
* Patients with metastatic disease.
* History of uncontrolled or labile hypertension, defined as blood pressure greater than 150/100mmHg (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.3.0 grade greater than or equal to 2), systolic blood pressure greater than 180 mm Hg if diastolic blood pressure less than 90 mm Hg, or diastolic blood pressure greater than 90 mm Hg, on at least 2 repeated determinations on separate days within 3 months prior to study enrollment. Patients who have medication controlled hypertension are eligible for the study.
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris or uncontrolled angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, clinically significant peripheral vascular disease (Grade II or greater).
* Psychiatric or neurologic illness that would limit compliance with study requirements.
* Patients with serious illness or medical condition.
* Active infection within 14 days before beginning treatment.
* Patients may not be receiving any other investigational agents.
* History of a malignancy in the last five years other than in situ carcinoma of the cervix, or non-melanomatous skin cancers.
* Patients must not be on therapeutic anticoagulation or chronic daily treatment with aspirin 325mg/day within 10 days prior to day 1 on study. Prophylactic anticoagulation during perioperative period is acceptable. Full dose aspirin post surgical resection is acceptable. Low dose aspirin 81mg/day and anticoagulation for line protection are allowed in the perioperative period and the adjuvant setting.
* Women who are breast feeding.
* History of stroke or transient ischemic attack within 6 months.
* History of pulmonary embolism, deep venous thrombosis or other thrombo-embolic event within 6 months prior to study.
* Patients with a history of severe hypersensitivity reaction to compounds of similar chemical or biologic composition to cisplatin, gemcitabine, bevacizumab, etoposide or other agents used in the study.
* History of a major surgical procedure, open biopsy, or a significant traumatic injury within 35 days prior to commencing treatment, or the anticipation of the need for a major surgical procedure during the course of the study prior to the predetermined date of tumor excision. Fine needle aspirations, core biopsies or mediastinoscopies within 7 days prior to commencing treatment.
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or tracheo-esophageal fistula.
* Non-healing wound or ulcer
* Evidence of coagulopathic disorder or hemorrhagic diathesis. International normalized ratio (INR) greater than 1.5.
* Patients with existing ototoxicity.
* Pregnancy (positive pregnancy test).
* Urine protein: creatinine ratio greater than or equal to 1.0 at screening.
* Patients known to be human immunodeficiency virus (HIV)-positive or have active hepatitis B/C (due to possible interaction between chemotherapy and highly active antiretroviral therapy (HAART) and antiviral medications used for treatment of active hepatitis B/C).
* Serious illness that may preclude adherence to the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- University Hospital for Lung Diseases, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre F, Grunenwald D, Pignon JP, Dujon A, Pujol JL, Brichon PY, Brouchet L, Quoix E, Westeel V, Le Chevalier T. Survival of patients with resected N2 non-small-cell lung cancer: evidence for a subclassification and implications. J Clin Oncol. 2000 Aug;18(16):2981-9. doi: 10.1200/JCO.2000.18.16.2981. PMID 10944131
- [Background] Vansteenkiste J, Betticher D, Eberhardt W, De Leyn P. Randomized controlled trial of resection versus radiotherapy after induction chemotherapy in stage IIIA-N2 non-small cell lung cancer. J Thorac Oncol. 2007 Aug;2(8):684-5. doi: 10.1097/JTO.0b013e31811f47ad. No abstract available. PMID 17762333
- [Background] Gilligan D, Nicolson M, Smith I, Groen H, Dalesio O, Goldstraw P, Hatton M, Hopwood P, Manegold C, Schramel F, Smit H, van Meerbeeck J, Nankivell M, Parmar M, Pugh C, Stephens R. Preoperative chemotherapy in patients with resectable non-small cell lung cancer: results of the MRC LU22/NVALT 2/EORTC 08012 multicentre randomised trial and update of systematic review. Lancet. 2007 Jun 9;369(9577):1929-37. doi: 10.1016/S0140-6736(07)60714-4. PMID 17544497
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0107.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage IIIA Lung Cancer Patients
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stage IIIA Lung Cancer Patients
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.76 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response
Description: Complete response is defined as a disappearance of all target lesions and was assessed by the RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
Time Frame: 25 weeks
Population: No goals were met because of low accrual for which the study was closed.
Arm/Group | Stage IIIA Lung Cancer Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the number of participants with adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. For the detailed list of adverse events see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 38 months
Measure: Count of Participants; unit: Participants
Arm/Group | Stage IIIA Lung Cancer Patients
Number analyzed (Participants) | 7
Participants | 7

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time between the first day of treatment to the day of disease progression. Progression will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: The time between the first day of treatment to the day of disease progression
Population: No goals were met because of low accrual for which the study was closed.
Arm/Group | Stage IIIA Lung Cancer Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Median Survival
Description: Median survival is the length of time a participant lives with disease following treatment.
Time Frame: Length of time a participant lives with disease following treatment
Population: No goals were met because of low accrual for which the study was closed.
Arm/Group | Stage IIIA Lung Cancer Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time between the first day of treatment to the day of death.
Time Frame: The time between the first day of treatment to the day of death
Population: No goals were met because of low accrual for which the study was closed.
Arm/Group | Stage IIIA Lung Cancer Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 38 months.
Arm/Group | Stage IIIA Lung Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage IIIA Lung Cancer Patients (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, embolism ) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage IIIA Lung Cancer Patients (N=7)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (5)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (4)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (10)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 1 (2)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Cardiac troponin I (cTnT) (Cardiac disorders) | 1 (2)
cholecystitis (Hepatobiliary disorders) | 1 (1)
Creatinine (Investigations) | 1 (3)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Investigations) | 2 (14)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Leukocytes (Investigations) | 6 (10)
Lymphopenia (Investigations) | 2 (5)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (10)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 (17)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (2)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (3)
Platelets (Investigations) | 4 (9)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No primary or secondary goals were met because of low accrual for which the study was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-12-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT00924209/Prot_SAP_000.pdf
  • Informed Consent Form (2009-01-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT00924209/ICF_001.pdf